CLINICAL TRIAL: NCT03345407
Title: A Phase IIb, Randomized (Stratified), Double-Blind (Sponsor Open), Parallel-Group, Placebo-Controlled, Dose-Finding Study of Nemiralisib (GSK2269557) Added to Standard of Care (SoC) Versus SoC Alone in Participants Diagnosed With an Acute Moderate or Severe Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Dose Finding Study of Nemiralisib (GSK2269557) in Subjects With an Acute Moderate or Severe Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unfavourable benefit:risk
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200879; 2017-001074-42 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Nemiralisib; Dose-Finding; GSK2269557; Acute Moderate or Severe Exacerbation of Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either nemiralisib (50-750 µg) or placebo in a parallel group.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind, sponsor- open study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- placebo once daily (Placebo Comparator): Eligible subjects will receive placebo ELLIPTA dry powder (blended with lactose) for oral inhalation once daily in the morning for 12 weeks. Albuterol (Salbutamol) MDI or nebules will also be provided to all subjects for use as rescue medication as needed.
  Interventions: Drug: Placebo ELLIPTA; Drug: Albuterol (Salbutamol) MDI or nebules; Drug: Standard of care therapy
- Nemiralisib 50 µg once daily (Experimental): Eligible subjects will receive nemiralisib ELLIPTA 50 µg dry powder (blended with lactose and magnesium stearate) for oral inhalation once daily in the morning for 12 weeks. Albuterol (Salbutamol) MDI or nebules will also be provided to all subjects for use as rescue medication as needed.
  Interventions: Drug: Nemiralisib ELLIPTA 50 µg; Drug: Albuterol (Salbutamol) MDI or nebules; Drug: Standard of care therapy
- Nemiralisib 100 µg once daily (Experimental): Eligible subjects will receive nemiralisib ELLIPTA 100 µg dry powder (blended with lactose and magnesium stearate) for oral inhalation once daily in the morning for 12 weeks. Albuterol (Salbutamol) MDI or nebules will also be provided to all subjects for use as rescue medication as needed.
  Interventions: Drug: Nemiralisib ELLIPTA 100 µg; Drug: Albuterol (Salbutamol) MDI or nebules; Drug: Standard of care therapy
- Nemiralisib 250 µg once daily (Experimental): Eligible subjects will receive nemiralisib ELLIPTA 250 µg dry powder (blended with lactose and magnesium stearate) for oral inhalation once daily in the morning for 12 weeks. Albuterol (Salbutamol) MDI or nebules will also be provided to all subjects for use as rescue medication as needed.
  Interventions: Drug: Nemiralisib ELLIPTA 250 µg; Drug: Albuterol (Salbutamol) MDI or nebules; Drug: Standard of care therapy
- Nemiralisib 500 µg once daily (Experimental): Eligible subjects will receive nemiralisib ELLIPTA 500 µg dry powder (blended with lactose and magnesium stearate) for oral inhalation once daily in the morning for 12 weeks. Albuterol (Salbutamol) MDI or nebules will also be provided to all subjects for use as rescue medication as needed.
  Interventions: Drug: Nemiralisib ELLIPTA 500 µg; Drug: Albuterol (Salbutamol) MDI or nebules; Drug: Standard of care therapy
- Nemiralisib 750 µg once daily (Experimental): Eligible subjects will receive nemiralisib ELLIPTA 750 µg dry powder (blended with lactose and magnesium stearate) for oral inhalation once daily in the morning for 12 weeks. Albuterol (Salbutamol) MDI or nebules will also be provided to all subjects for use as rescue medication as needed.
  Interventions: Drug: Nemiralisib ELLIPTA 750 µg; Drug: Albuterol (Salbutamol) MDI or nebules; Drug: Standard of care therapy

INTERVENTIONS:
Drug: Placebo ELLIPTA — Placebo will be administered via oral inhalation route once daily in the morning.
  Arms: placebo once daily
Drug: Nemiralisib ELLIPTA 50 µg — Nemiralisib is a potent and highly selective inhaled PI3Kd inhibitor being developed as an anti-inflammatory for the treatment of inflammatory airways disease. Nemiralisib 50 µg will be administered as a dry powder inhaler via oral inhalation route. In addition, subjects will receive SOC therapy for the index acute moderate or severe exacerbation of COPD.
  Arms: Nemiralisib 50 µg once daily
Drug: Nemiralisib ELLIPTA 100 µg — Nemiralisib is a potent and highly selective inhaled PI3Kd inhibitor being developed as an anti-inflammatory for the treatment of inflammatory airways disease. Nemiralisib 100 µg will be administered as a dry powder inhaler via oral inhalation route. In addition, subjects will receive SOC therapy for the index acute moderate or severe exacerbation of COPD.
  Arms: Nemiralisib 100 µg once daily
Drug: Nemiralisib ELLIPTA 250 µg — Nemiralisib is a potent and highly selective inhaled PI3Kd inhibitor being developed as an anti-inflammatory for the treatment of inflammatory airways disease. Nemiralisib 250 µg will be administered as a dry powder inhaler via oral inhalation route. In addition, subjects will receive SOC therapy for the index acute moderate or severe exacerbation of COPD.
  Arms: Nemiralisib 250 µg once daily
Drug: Nemiralisib ELLIPTA 500 µg — Nemiralisib is a potent and highly selective inhaled PI3Kd inhibitor being developed as an anti-inflammatory for the treatment of inflammatory airways disease. Nemiralisib 500 µg will be administered as a dry powder inhaler via oral inhalation route. In addition, subjects will receive SOC therapy for the index acute moderate or severe exacerbation of COPD.
  Arms: Nemiralisib 500 µg once daily
Drug: Nemiralisib ELLIPTA 750 µg — Nemiralisib is a potent and highly selective inhaled PI3Kd inhibitor being developed as an anti-inflammatory for the treatment of inflammatory airways disease. Nemiralisib 750 µg will be administered as a dry powder inhaler via oral inhalation route. In addition, subjects will receive SOC therapy for the index acute moderate or severe exacerbation of COPD.
  Arms: Nemiralisib 750 µg once daily
Drug: Albuterol (Salbutamol) MDI or nebules — Albuterol (Salbutamol) MDI or nebules will be provided to all subjects as a rescue medication.
Drug: Standard of care therapy — SoC therapy for the index exacerbation is defined as treatment with oral/systemic corticosteroid (prednisone 40 mg/day or equivalent) for 5 days and antibiotic for 7 days. Subjects will receive SoC as prescribed by the Investigator or medically qualified designee. The dose and/or duration of prednisone and/or the antibiotic can be modified according to the Investigator's/medically qualified designee's judgment or according to local country/institution practice.

SUMMARY:
Nemiralisib is being developed as an anti-inflammatory drug for the treatment of inflammatory airways disease. This study is designed to assess the dose response, efficacy, safety, and pharmacokinetics of nemiralisib across a range of doses [up to 750 micrograms (µg)] compared with placebo. The study consists of a Screening Period, a 12-Week Treatment Period and a 12-Week Post-Treatment Follow-Up Period. Approximately 1,250 subjects with an acute moderate or severe exacerbation of COPD requiring standard of care (SoC) therapy will be randomized in this double-blind study. Subjects will be randomized to receive different doses of nemiralisib or placebo via ELLIPTA® inhaler. The total duration of study participation is approximately 6 months (170 days). ELLIPTA is the registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 80 years of age, inclusive, at Screening (Visit 1).
* An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society [ global initiative for chronic obstructive lung disease (GOLD), 2017] as follows: "Chronic obstructive pulmonary disease is a common, preventable and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases."
* Current or former cigarette smoker with a history of cigarette smoking of >=10 pack-years. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Screening (Visit 1). Number of pack years = (number of cigarettes per day / 20) x number of years smoked).
* Acute exacerbation of COPD requiring an escalation in therapy to include oral/systemic corticosteroid(s) (prednisone 40 mg/day or equivalent) for 5 days and antibiotic(s) for 7 days; the dose and/or duration of prednisone (40 mg/day or equivalent) and/or the antibiotic can be modified according to the Investigator's/medically qualified designee's judgment or according to local country/institution practice. Acute exacerbation to be confirmed by an experienced physician and to represent a recent worsening of at least two major and one minor symptoms, one major and two minor symptoms, or all 3 major symptoms. Major symptoms include subjective increase in dyspnea, increase in sputum volume or change in sputum color. Minor symptoms include increased cough, increased wheeze, sore throat, colds or fever (oral temperature >37.5 degree Celsius) without other cause.
* Body weight >=45 kilogram (kg) and body mass index (BMI) within the range 16 - 35 kg per meter square (kg/m^2) (inclusive)
* Male and female subjects are eligible to participate in the study. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the 12-Week Double-Blind Treatment Period and for at least 5 half-lives (10 days) after the last of double-blind study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Current diagnosis of asthma, according to the Global Initiative for Asthma (GINA, 2017). Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD.
* Potential of hydrogen (pH) < 7.30 or the need for invasive mechanical ventilation.
* Moderate/severe exacerbation of COPD for which SoC was started >48 hours since diagnosis.
* A chest X-ray [or computed tomography (CT) scan] that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray (or CT scan) must be taken at Screening (Visit 1). For sites in Germany: if a chest X-ray (or CT scan) within 1 year of Screening (Visit 1) is not available, approval to conduct a diagnostic chest X-ray (CT scan) will need to be obtained from the Federal Office for Radiation Protection (BfS).
* Clinically significant pneumonia, identified by chest X-ray (CT scan) at Screening.
* A diagnosis of alpha 1-antitrypsin deficiency as the underlying cause of COPD, active tuberculosis, lung cancer, clinically overt bronchiectasis (Note: focal bronchiectasis is not exclusionary), sarcoidosis, pulmonary fibrosis (Note: focal fibrotic pulmonary lesions are not exclusionary), primary pulmonary hypertension, interstitial lung diseases,or any other respiratory condition that might, in the opinion of the investigator, compromise the safety of the subject or affect the interpretation of the results.
* A history or current evidence of clinically significant and unstable disease such as cardiovascular (e.g., subjects requiring implanted cardioverter defibrillator [ICD], pacemaker requiring a rate set >60 beats per minute (bpm), uncontrolled hypertension, New Your Heart Association Class IV [NYHA, 1994], known left ventricular ejection fraction <30 percent) neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease), peptic ulcer disease, or hematological abnormalities. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study. (Note: subjects with adequately treated and well controlled concurrent medical conditions (e.g. hypertension or noninsulin-dependent diabetes mellitus [NIDDM]) are permitted to be entered into the study).
* Having undergone lung volume reduction surgery or lung resection for any other reason e.g. lung carcinoma
* Liver diseases including ALT>2x upper limit of normal (ULN); Total bilirubin >1.5xULN (Isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent); current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones); Presence of hepatitis B surface antigen (HBsAg) at Screening or within 3 months prior to first dose of study treatment; Positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of study treatment.
* Positive hepatitis C ribonucleic acid (RNA) test result at Screening or within 3 months prior to first dose of study treatment.
* Carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin are not excluded if the subject has been considered cured within 5 years since diagnosis.
* History of allergy or hypersensitivity to any of the study medications [e.g. beta-agonists, Phosphoinositide 3-Kinase Delta (PI3Kd) inhibitors] or components of the inhalation powder (e.g., lactose). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the investigator, contraindicates the subject's participation are excluded.
* Strong inhibitors of cytochrome P450 3A4 (CYP3A4) including antiretrovirals including protease inhibitors; Oral antifungal treatments such as ketoconazole and itraconazole. It is recommended that posaconazole is used as the oral antifungal treatment of choice. Short courses of up to 14 days are allowed for fluconazole and voriconazole, but chronic administrations are not permitted; Antibiotics such as telithromycin and troleandomycin (macrolide). It is recommended that azithromycin is used as the macrolide antibiotic of choice. Short courses up to 14 days are allowed for mibefradil (calcium channel blocker), erythromycin and clarithromycin (including intravenous clarithromycin) but chronic administrations are not permitted; Anti-epileptic treatments; and anti-tuberculosis therapy. These medications must all have been stopped at least 14 days prior to first dose of study treatment. Use of sensitive narrow therapeutic index CYP3A4 substrates including alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus and tacrolimus; Intravenous theophylline will be allowed but only under strict therapeutic drug monitoring for signs of theophylline toxicity as a result of co-administration with nemiralisib; Subjects may be recruited into the study already under treatment with theophylline or started on theophylline following the start of treatment and before the end of 14 days post last dose.
* Chronic treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for >15 hours a day. Oxygen prn use (<=15 hours per day) is not exclusionary. Oxygen use during an exacerbation is permitted.
* Chronic treatment with anti-Tumor Necrosis Factor (anti-TNF), anti-Interleukin-1 (anti-IL1), or any other immunosuppressive therapy within 60 days prior to the first dose of double-blind study treatment.
* Clinically significant sleep apnea that requires the use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) for > 48 hours.
* Any other investigational treatment within the following time periods prior to the first dose of double-blind study treatment in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product, whichever is longer. Note: subjects who participated in a previously completed study and/or were withdrawn from an ongoing study that included/includes nemiralisib are excluded from participating in this study.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dose of double-blind study treatment in the current study.
* A clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the exclusion criteria, outside of the reference range for the population being studied may be included if the Investigator [in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required] documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Abnormal, clinically significant ECG finding (e.g. myocardial Infarction or demonstrating a clinically significant arrhythmia requiring treatment) at Screening (Visit 1) or upon repeat prior to randomization.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >480 milliseconds (msec) for subjects with or without Bundle Branch Block, based on single QTcF value.
* A positive test for human immunodeficiency virus (HIV) antibody at Screening.
* Known or suspected history of alcohol or drug abuse within the last 2 years.
* History of regular alcohol consumption defined as an average weekly intake of >28 units for males or >21 units for females within 6 months of Screening (Visit 1). One unit is equivalent to 8 grams of alcohol: a half-pint [approximately 240 milliliter (mL)] of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (145):
- United States (20):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (9):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santo Tomé, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (6):
  - GSK Investigational Site, Gosford, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Woodville South, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- France (5):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (15):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Italy (8):
  - GSK Investigational Site, Reggio Emilia, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Messina, Sicily
  - GSK Investigational Site, Negrar, Veneto
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
- Netherlands (9):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zwolle
- Poland (9):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Oława
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Sosnowiec
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Tarnów
- Romania (8):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Comuna Alexandru Cel Bun
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (15):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Veliky Novgorod
  - GSK Investigational Site, Voronezh
- South Korea (5):
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju-si, Jeollabuk-do
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (15):
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Elda (Alicante)
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Orihuela (Alicante)
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pama de Mallorca
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
- United Kingdom (9):
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Wishaw, Lanarkshire
  - GSK Investigational Site, Blackburn
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Edgbaston
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20850

REFERENCES:
- [Background] Fahy WA, Homayoun-Valiani F, Cahn A, Robertson J, Templeton A, Meeraus WH, Wilson R, Lowings M, Marotti M, West SL, Tabberer M, Hessel EM. Nemiralisib in Patients with an Acute Exacerbation of COPD: Placebo-Controlled, Dose-Ranging Study. Int J Chron Obstruct Pulmon Dis. 2021 Jun 3;16:1637-1646. doi: 10.2147/COPD.S309320. eCollection 2021. PMID 34113095

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIb, multicenter, randomized, stratified, double-blind (sponsor open), placebo controlled parallel-group study in participants who presented with an acute moderate or severe exacerbation of chronic obstructive pulmonary disease (COPD) requiring Standard of Care (SoC).
Pre-assignment Details: A total of 943 participants were randomized, and 938 participants who received at least one dose of study treatment were included in the modified intent to treat (MITT) Population. The study included participants enrolled from 16 countries.
Groups:
- Placebo: Participants were administered a single oral inhalation of placebo via ELLIPTA dry powder inhaler (DPI) once daily in the morning for 12 weeks. Albuterol (salbutamol) metered-dose inhaler (MDI) or nebules were also provided to all participants as rescue medication.
- Nemiralisib 12.5 mcg: Participants were administered a single oral inhalation of 12.5 micrograms (mcg) nemiralisib via ELLIPTA DPI once daily in the morning for 12 weeks. Albuterol (salbutamol) MDI or nebules were also provided to all participants as rescue medication.
- Nemiralisib 50 mcg: Participants were administered a single oral inhalation of 50 mcg nemiralisib via ELLIPTA DPI once daily in the morning for 12 weeks. Albuterol (salbutamol) MDI or nebules were also provided to all participants as rescue medication.
- Nemiralisib 100 mcg: Participants were administered a single oral inhalation of 100 mcg nemiralisib via ELLIPTA DPI once daily in the morning for 12 weeks. Albuterol (salbutamol) MDI or nebules were also provided to all participants as rescue medication.
- Nemiralisib 250 mcg: Participants were administered a single oral inhalation of 250 mcg nemiralisib via ELLIPTA DPI once daily in the morning for 12 weeks. Albuterol (salbutamol) MDI or nebules were also provided to all participants as rescue medication.
- Nemiralisib 500 mcg: Participants were administered a single oral inhalation of 500 mcg nemiralisib via ELLIPTA DPI once daily in the morning for 12 weeks. Albuterol (salbutamol) MDI or nebules were also provided to all participants as rescue medication.
- Nemiralisib 750 mcg: Participants were administered a single oral inhalation of 750 mcg nemiralisib via ELLIPTA DPI once daily in the morning for 12 weeks. Albuterol (salbutamol) MDI or nebules were also provided to all participants as rescue medication.
Period: Overall Study
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Started | 276 | 22 | 91 | 92 | 90 | 89 | 278
Completed | 244 | 19 | 79 | 81 | 75 | 73 | 233
Not Completed | 32 | 3 | 12 | 11 | 15 | 16 | 45
Not completed — Withdrawal by Subject | 11 | 1 | 5 | 6 | 3 | 6 | 16
Not completed — Physician Decision | 3 | 1 | 0 | 0 | 1 | 2 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 1 | 2 | 3
Not completed — Protocol-defined stopping criteria | 9 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Lack of Efficacy | 1 | 1 | 1 | 1 | 1 | 0 | 3
Not completed — Adverse Event | 4 | 0 | 5 | 4 | 6 | 5 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg | Total
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278 | 938
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (7.94) | 67.8 (7.20) | 63.1 (7.61) | 65.1 (7.43) | 66.0 (6.94) | 64.9 (8.04) | 64.8 (7.61) | 65.0 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 6 | 35 | 29 | 31 | 22 | 100 | 309
  Male | 190 | 16 | 56 | 63 | 59 | 67 | 178 | 629
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 1 | 2 | 2 | 6 | 15
  Asian-East Asian Heritage | 18 | 4 | 7 | 2 | 9 | 7 | 19 | 66
  Asian-South East Asian Heritage | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 4
  Black or African American | 2 | 1 | 2 | 1 | 0 | 2 | 6 | 14
  White-Arabic/North African Heritage | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4
  White-White Caucasian/European Heritage | 252 | 17 | 79 | 86 | 79 | 76 | 246 | 835

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Visit Trough Forced Expiratory Volume in One Second (FEV1) at Day 84 Measured Post Bronchodilator
Description: FEV1 is maximal amount of air exhaled forcefully from lungs in 1 second. Post-bronchodilator FEV1 was conducted approximately 10-30 minutes after participant was administered 4 inhalations of albuterol (salbutamol) via MDI using spacer/valved-holding chamber or via one nebulized treatment. Post-bronchodilator Baseline FEV1 is latest FEV1 measured prior to first dose of study treatment and post-bronchodilator. Change from Baseline in clinic visit trough FEV1 at Day 84 measured post-bronchodilator is FEV1 measured prior to dosing and post-bronchodilator on Day 84 minus post-bronchodilator Baseline FEV1. Bayesian repeated measure model adjusted for Baseline by visit interaction, treatment by visit interaction, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in previous 12 months and gender was used. Posterior adjusted median change from Baseline and 95% highest posterior density (HPD) credible interval (CrI) was presented.
Time Frame: Baseline and Day 84
Population: MITT Population consisted of all randomized participants who received at least 1 dose of study treatment.. Only those participants with data available at the specified data points were analyzed.
Measure: Median (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 215 | 16 | 72 | 75 | 69 | 58 | 216
Liters | 0.052 [0.018 to 0.091] | 0.031 [-0.090 to 0.149] | 0.026 [-0.036 to 0.084] | 0.014 [-0.044 to 0.073] | 0.058 [-0.002 to 0.118] | 0.049 [-0.017 to 0.113] | 0.049 [0.012 to 0.086]
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = -0.022, 95% CI 2-sided [-0.143 to 0.103] — Treatment comparison (posterior adjusted median difference and 95% HPD CrI) of Nemiralisib 12.5 mcg and placebo for Day 84 change from Baseline FEV1 measured post-bronchodilator has been presented
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = -0.027, 95% CI 2-sided [-0.098 to 0.036] — Treatment comparison (posterior adjusted median difference and 95% HPD CrI) of Nemiralisib 50 mcg and placebo for Day 84 change from Baseline FEV1 measured post-bronchodilator has been presented
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = -0.038, 95% CI 2-sided [-0.102 to 0.028] — Treatment comparison (posterior adjusted median difference and 95% HPD CrI) of Nemiralisib 100 mcg and placebo for Day 84 change from Baseline FEV1 measured post-bronchodilator has been presented
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = 0.005, 95% CI 2-sided [-0.064 to 0.071] — Treatment comparison (posterior adjusted median difference and 95% HPD CrI) of Nemiralisib 250 mcg and placebo for Day 84 change from Baseline FEV1 measured post-bronchodilator has been presented
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjusted median difference = -0.003, 95% CI 2-sided [-0.075 to 0.061] — Treatment comparison (posterior adjusted median difference and 95% HPD CrI) of Nemiralisib 500 mcg and placebo for Day 84 change from Baseline FEV1 measured post-bronchodilator has been presented
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = -0.004, 95% CI 2-sided [-0.051 to 0.042] — Treatment comparison (posterior adjusted median difference and 95% HPD CrI) of Nemiralisib 750 mcg and placebo for Day 84 change from Baseline FEV1 measured post-bronchodilator has been presented

2. Secondary Outcome: Rate of Moderate and Severe Exacerbations Over 12-week Treatment Period
Description: Moderate COPD exacerbations are defined as worsening symptoms of COPD treated with short-acting bronchodilators (SABDs) plus antibiotics and/or oral/systemic corticosteroids. Severe COPD exacerbations are defined as worsening symptoms of COPD that require hospitalization or visit to the emergency room. Severe exacerbation may also be associated with acute respiratory failure. Rate of exacerbations was analyzed using Bayesian Poisson model adjusting for length of on-treatment follow-up, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in the previous 12 months and gender. Posterior median exacerbation rate and 95% HPD CrI has been presented.
Time Frame: Up to Week 12
Population: MITT Population.
Measure: Median (95% Confidence Interval); unit: No.of exacerbation per 84 Days
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
No.of exacerbation per 84 Days | 0.31 [0.25 to 0.39] | NA [NA to NA] — The participants randomized to Nemiralisib 12.5 mcg were excluded from this analysis due to insufficient participants with data. | 0.29 [0.20 to 0.39] | 0.28 [0.20 to 0.38] | 0.32 [0.23 to 0.43] | 0.20 [0.13 to 0.29] | 0.36 [0.29 to 0.43]
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median exacerbation rate ratio = 0.92, 95% CI 2-sided [0.60 to 1.40] — Treatment comparison (posterior median exacerbation rate ratio and 95% HPD CrI) of Nemiralisib 50 mcg and placebo for moderate/severe exacerbations has been presented
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median exacerbation rate ratio = 0.89, 95% CI 2-sided [0.57 to 1.35] — Treatment comparison (posterior median exacerbation rate ratio and 95% HPD CrI) of Nemiralisib 100 mcg and placebo for moderate/severe exacerbations has been presented
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median exacerbation rate ratio = 1.01, 95% CI 2-sided [0.65 to 1.50] — Treatment comparison (posterior median exacerbation rate ratio and 95% HPD CrI) of Nemiralisib 250 mcg and placebo for moderate/severe exacerbations has been presented
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median exacerbation rate ratio = 0.63, 95% CI 2-sided [0.37 to 1.02] — Treatment comparison (posterior median exacerbation rate ratio and 95% HPD CrI) of Nemiralisib 500 mcg and placebo for moderate/severe exacerbations has been presented
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median exacerbation rate ratio = 1.13, 95% CI 2-sided [0.85 to 1.52] — Treatment comparison (posterior median exacerbation rate ratio and 95% HPD CrI) of Nemiralisib 750 mcg and placebo for moderate/severe exacerbations has been presented

3. Secondary Outcome: Number of Participants With Time to Next Moderate/Severe Exacerbation Following Index Exacerbation
Description: Number of participants with time to next (on-treatment) moderate/severe exacerbation following index exacerbation during the 12-Week Treatment Period was defined as time from the date of randomization until the date of onset of the first moderate/severe exacerbation whilst on study treatment. Participants who did not have an exacerbation whilst on study treatment were censored at the date of their last dose of study treatment. Time to next exacerbation was analyzed using a Bayesian Cox proportional hazards model adjusting for treatment group, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in the previous 12 months and gender.
Time Frame: Up to Week 12
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants | 72 | 3 | 24 | 25 | 26 | 15 | 80
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median hazard ratio = 0.455, 95% CI 2-sided [0.054 to 1.103] — Treatment comparison (Hazard Ratio and 95% HPD CrI) of Nemiralisib 12.5 mcg and placebo for time to next moderate/severe exacerbations has been presented
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median hazard ratio = 0.991, 95% CI 2-sided [0.580 to 1.500] — Treatment comparison (Hazard Ratio and 95% HPD CrI) of Nemiralisib 50 mcg and placebo for time to next moderate/severe exacerbations has been presented
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median hazard ratio = 0.975, 95% CI 2-sided [0.581 to 1.467] — Treatment comparison (Hazard Ratio and 95% HPD CrI) of Nemiralisib 100 mcg and placebo for time to next moderate/severe exacerbations has been presented
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median hazard ratio = 1.132, 95% CI 2-sided [0.682 to 1.709] — Treatment comparison (Hazard Ratio and 95% HPD CrI) of Nemiralisib 250 mcg and placebo for time to next moderate/severe exacerbations has been presented
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median hazard ratio = 0.556, 95% CI 2-sided [0.268 to 0.902] — Treatment comparison (Hazard Ratio and 95% HPD CrI) of Nemiralisib 500 mcg and placebo for time to next moderate/severe exacerbations has been presented
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median hazard ratio = 1.149, 95% CI 2-sided [0.800 to 1.539] — Treatment comparison (Hazard Ratio and 95% HPD CrI) of Nemiralisib 750 mcg and placebo for time to next moderate/severe exacerbations has been presented

4. Secondary Outcome: Change From Baseline in Clinic Visit Trough FEV1 Measured Pre and Post-bronchodilator
Description: Pulmonary function was measured by FEV1, defined as maximal amount of air exhaled forcefully from the lungs in 1 second. Post-bronchodilator FEV1 was conducted approximately 10-30 minutes after participant was administered with 4 inhalations of albuterol via MDI using a spacer/valved-holding chamber or via 1 nebulized treatment. Pre-bronchodilator and post-bronchodilator Baseline FEV1 is latest FEV1 measured prior to first dose of study treatment and pre-bronchodilator and post-bronchodilator, respectively. Change from Baseline in clinic visit trough FEV1 at Days 14, 28, 56 and 84 measured pre-bronchodilator is defined as FEV1 measured prior to dosing and pre-bronchodilator on Days 14, 28, 56 and 84 minus pre-bronchodilator Baseline FEV1.
Time Frame: Baseline and Days 14, 28, 56 (pre and post bronchodilaor), 84 (pre-bronchodilator) and at hospital discharge (maximum 24 Weeks)
Population: MITT Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Liters
  Day 14, Pre, n=240, 20, 85, 83, 76, 76, 238: number analyzed (Participants) | 240 | 20 | 85 | 83 | 76 | 76 | 238
  Day 14, Pre, n=240, 20, 85, 83, 76, 76, 238 | 0.008 (0.2729) | 0.100 (0.2511) | -0.021 (0.2657) | -0.013 (0.2509) | 0.053 (0.2958) | 0.041 (0.2738) | 0.023 (0.2561)
  Day 14, Post, n=248, 20, 86, 83, 77, 78, 241: number analyzed (Participants) | 248 | 20 | 86 | 83 | 77 | 78 | 241
  Day 14, Post, n=248, 20, 86, 83, 77, 78, 241 | 0.034 (0.2707) | 0.075 (0.2425) | 0.010 (0.2168) | -0.050 (0.2477) | 0.054 (0.2983) | 0.073 (0.2655) | 0.044 (0.2216)
  Day 28, Pre, n=239, 20, 82, 79, 75, 71, 232: number analyzed (Participants) | 239 | 20 | 82 | 79 | 75 | 71 | 232
  Day 28, Pre, n=239, 20, 82, 79, 75, 71, 232 | 0.017 (0.2585) | 0.081 (0.2661) | -0.034 (0.2875) | -0.010 (0.2333) | 0.064 (0.2592) | 0.016 (0.2713) | 0.020 (0.2512)
  Day 28, Post, n=245, 19, 83, 81, 76, 72, 232: number analyzed (Participants) | 245 | 19 | 83 | 81 | 76 | 72 | 232
  Day 28, Post, n=245, 19, 83, 81, 76, 72, 232 | 0.036 (0.2647) | 0.059 (0.2575) | 0.004 (0.2183) | -0.034 (0.2401) | 0.049 (0.2639) | 0.027 (0.2369) | 0.029 (0.2307)
  Day 56, Pre, n=230, 20, 78, 76, 73, 67, 224: number analyzed (Participants) | 230 | 20 | 78 | 76 | 73 | 67 | 224
  Day 56, Pre, n=230, 20, 78, 76, 73, 67, 224 | 0.005 (0.2295) | -0.006 (0.2636) | -0.024 (0.3210) | 0.011 (0.2415) | 0.022 (0.2522) | -0.004 (0.2233) | -0.001 (0.2858)
  Day 56, Post, n=237, 19, 78, 77, 74, 69, 224: number analyzed (Participants) | 237 | 19 | 78 | 77 | 74 | 69 | 224
  Day 56, Post, n=237, 19, 78, 77, 74, 69, 224 | 0.020 (0.2614) | -0.002 (0.2252) | -0.012 (0.2524) | 0.004 (0.2373) | 0.026 (0.2556) | -0.011 (0.2260) | 0.011 (0.2470)
  Day 84, Pre, n=210, 17, 71, 73, 66, 58, 212: number analyzed (Participants) | 210 | 17 | 71 | 73 | 66 | 58 | 212
  Day 84, Pre, n=210, 17, 71, 73, 66, 58, 212 | 0.000 (0.2566) | 0.003 (0.2232) | -0.049 (0.2549) | 0.005 (0.2668) | 0.015 (0.2739) | 0.007 (0.2461) | 0.010 (0.2829)
  Hospital discharge, Pre, n=23, 2, 8, 8, 7, 3, 22: number analyzed (Participants) | 23 | 2 | 8 | 8 | 7 | 3 | 22
  Hospital discharge, Pre, n=23, 2, 8, 8, 7, 3, 22 | 0.071 (0.1586) | 0.168 (0.2652) | 0.108 (0.3888) | 0.056 (0.1782) | 0.052 (0.3481) | 0.162 (0.1426) | 0.075 (0.1974)
  Hospital discharge, Post, n=8, 2, 1, 1, 1, 0, 6: number analyzed (Participants) | 8 | 2 | 1 | 1 | 1 | 0 | 6
  Hospital discharge, Post, n=8, 2, 1, 1, 1, 0, 6 | 0.134 (0.1514) | 0.153 (0.0933) | 0.083 (NA) — Not applicable (NA) indicates standard deviation could not be calculated as single participant was analyzed. | -0.076 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. | 0.094 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. |  | -0.006 (0.1079)

5. Secondary Outcome: Change From Hospital Discharge in Clinic Visit Trough FEV1 Measured Pre and Post-bronchodilator
Description: Pulmonary function was measured by FEV1, defined as maximal amount of air exhaled forcefully from the lungs in 1 second. Post-bronchodilator FEV1 was conducted approximately 10 to 30 minutes after participant was administered with 4 inhalations of albuterol via MDI using a spacer/valved-holding chamber or via 1 nebulized treatment. Pre-bronchodilator and post-bronchodilator Baseline FEV1 is defined as latest FEV1 measured prior to first dose of study treatment and pre-bronchodilator and post-bronchodilator, respectively. Change from hospital discharge in clinic visit trough FEV1 at Days 14, 28, 56 and 84 measured pre- and post-bronchodilator is defined as FEV1 measured prior to dosing and pre- and post-bronchodilator on Days 14, 28, 56 and 84 minus pre and post-bronchodilator Baseline FEV1.
Time Frame: Baseline and pre- and post-bronchodilator on Days 14, 28, 56 and 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Liters
  Day 14, Pre, n=20, 2, 8, 8, 6, 4, 20: number analyzed (Participants) | 20 | 2 | 8 | 8 | 6 | 4 | 20
  Day 14, Pre, n=20, 2, 8, 8, 6, 4, 20 | 0.082 (0.2783) | 0.355 (0.4207) | 0.069 (0.3012) | -0.049 (0.1882) | -0.069 (0.4905) | 0.173 (0.5137) | 0.002 (0.2343)
  Day 14, Post, n=5, 2, 1, 1, 1, 0, 5: number analyzed (Participants) | 5 | 2 | 1 | 1 | 1 | 0 | 5
  Day 14, Post, n=5, 2, 1, 1, 1, 0, 5 | 0.056 (0.3372) | 0.431 (0.5190) | 0.119 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. | 0.310 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. | -0.305 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. |  | -0.021 (0.1326)
  Day 28, Pre, n=37, 2, 14, 8, 10, 9, 37: number analyzed (Participants) | 37 | 2 | 14 | 8 | 10 | 9 | 37
  Day 28, Pre, n=37, 2, 14, 8, 10, 9, 37 | 0.026 (0.2691) | 0.261 (0.5204) | 0.012 (0.2910) | -0.085 (0.2072) | 0.012 (0.4020) | 0.030 (0.4029) | -0.046 (0.2639)
  Day 28, Post, n=22, 2, 8, 1, 4, 4, 22: number analyzed (Participants) | 22 | 2 | 8 | 1 | 4 | 4 | 22
  Day 28, Post, n=22, 2, 8, 1, 4, 4, 22 | 0.034 (0.2779) | 0.334 (0.5614) | 0.130 (0.2327) | 0.130 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. | 0.009 (0.2006) | 0.007 (0.3237) | -0.094 (0.2293)
  Day 56, Pre, n=37, 2, 14, 8, 9, 10, 36: number analyzed (Participants) | 37 | 2 | 14 | 8 | 9 | 10 | 36
  Day 56, Pre, n=37, 2, 14, 8, 9, 10, 36 | 0.019 (0.2282) | 0.106 (0.6138) | 0.019 (0.3509) | 0.014 (0.1938) | -0.074 (0.3847) | -0.042 (0.1840) | -0.054 (0.2942)
  Day 56, Post, n=22, 2, 7, 1, 4, 5, 21: number analyzed (Participants) | 22 | 2 | 7 | 1 | 4 | 5 | 21
  Day 56, Post, n=22, 2, 7, 1, 4, 5, 21 | -0.014 (0.2896) | 0.139 (0.6838) | 0.042 (0.3068) | 0.098 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. | -0.056 (0.3572) | -0.072 (0.1490) | -0.135 (0.2410)
  Day 84, Pre, n=37, 2, 12, 8, 7, 10, 35: number analyzed (Participants) | 37 | 2 | 12 | 8 | 7 | 10 | 35
  Day 84, Pre, n=37, 2, 12, 8, 7, 10, 35 | 0.007 (0.2741) | -0.027 (0.4554) | 0.121 (0.2770) | -0.081 (0.1738) | -0.072 (0.4391) | 0.043 (0.2511) | -0.062 (0.2816)
  Day 84, Post, n=22, 2, 6, 1, 4, 5, 22: number analyzed (Participants) | 22 | 2 | 6 | 1 | 4 | 5 | 22
  Day 84, Post, n=22, 2, 6, 1, 4, 5, 22 | -0.039 (0.2610) | 0.133 (0.5162) | 0.037 (0.3341) | 0.108 (NA) — NA indicates standard deviation could not be calculated as single participant was analyzed. | 0.021 (0.3151) | 0.006 (0.2180) | -0.106 (0.2956)

6. Secondary Outcome: Percentage of Participants Achieving the Exacerbations of Chronic Pulmonary Disease Tool (EXACT) Definition of Recovery From the Index Exacerbation
Description: EXACT patient-reported outcome (EXACT-PRO), 14-item instrument to capture occurrence, frequency, severity, and duration of exacerbations using an electronic diary (eDiary). Total score ranges from 0-100, higher score indicates more severe condition. Participants were required to complete EXACT-PRO every evening; however, on the day of randomization it was to be completed in the morning. Response was decrease in rolling average EXACT Total Score >=9 points from maximum observed value, sustained for >=7 days, with first of 7 days defined as recovery day. Analysis was performed using Bayesian Cox proportional hazards model adjusting for treatment group, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in previous 12 months and gender.
Time Frame: Days 14, 28, 56 and 84
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Percentage of participants
  Day 14 | 29 | 27 | 37 | 29 | 28 | 24 | 32
  Day 28 | 40 | 41 | 52 | 43 | 42 | 27 | 42
  Day 56 | 49 | 45 | 59 | 52 | 50 | 31 | 50
  Day 84 | 51 | 50 | 59 | 54 | 50 | 37 | 54
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 1.01, 95% CI 2-sided [0.21 to 2.30] — Treatment comparison between placebo and nemiralisib 12.5 mcg at Day 14 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.37, 95% CI 2-sided [0.76 to 2.17] — Treatment comparison between placebo and nemiralisib 50 mcg at Day 14 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 0.99, 95% CI 2-sided [0.54 to 1.61] — Treatment comparison between placebo and nemiralisib 100 mcg at Day 14 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 0.94, 95% CI 2-sided [0.50 to 1.49] — Treatment comparison between placebo and nemiralisib 250 mcg at Day 14 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.75, 95% CI 2-sided [0.38 to 1.25] — Treatment comparison between placebo and nemiralisib 500 mcg at Day 14 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 1.16, 95% CI 2-sided [0.77 to 1.63] — Treatment comparison between placebo and nemiralisib 750 mcg at Day 14 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 7: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 1.21, 95% CI 2-sided [0.36 to 2.69] — Treatment comparison between placebo and nemiralisib 12.5 mcg at Day 28 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 8: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.53, 95% CI 2-sided [0.82 to 2.33] — Treatment comparison between placebo and nemiralisib 50 mcg at Day 28 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 9: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.16, 95% CI 2-sided [0.67 to 1.79] — Treatment comparison between placebo and nemiralisib 100 mcg at Day 28 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 10: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.12, 95% CI 2-sided [0.63 to 1.74] — Treatment comparison between placebo and nemiralisib 250 mcg at Day 28 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 11: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.55, 95% CI 2-sided [0.28 to 0.88] — Treatment comparison between placebo and nemiralisib 500 mcg at Day 28 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 12: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 1.08, 95% CI 2-sided [0.72 to 1.49] — Treatment comparison between placebo and nemiralisib 750 mcg at Day 28 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 13: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 1.00, 95% CI 2-sided [0.30 to 2.17] — Treatment comparison between placebo and nemiralisib 12.5 mcg at Day 56 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 14: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.46, 95% CI 2-sided [0.84 to 2.27] — Treatment comparison between placebo and nemiralisib 50 mcg at Day 56 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 15: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.15, 95% CI 2-sided [0.65 to 1.78] — Treatment comparison between placebo and nemiralisib 100 mcg at Day 56 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 16: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.09, 95% CI 2-sided [0.62 to 1.67] — Treatment comparison between placebo and nemiralisib 250 mcg at Day 56 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 17: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.49, 95% CI 2-sided [0.26 to 0.77] — Treatment comparison between placebo and nemiralisib 500 mcg at Day 56 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 18: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 1.04, 95% CI 2-sided [0.71 to 1.42] — Treatment comparison between placebo and nemiralisib 750 mcg at Day 56 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 19: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 1.08, 95% CI 2-sided [0.32 to 2.38] — Treatment comparison between placebo and nemiralisib 12.5 mcg at Day 84 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 20: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.29, 95% CI 2-sided [0.70 to 2.00] — Treatment comparison between placebo and nemiralisib 50 mcg at Day 84 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 21: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.12, 95% CI 2-sided [0.63 to 1.71] — Treatment comparison between placebo and nemiralisib 100 mcg at Day 84 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 22: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 0.95, 95% CI 2-sided [0.55 to 1.48] — Treatment comparison between placebo and nemiralisib 250 mcg at Day 84 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 23: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.56, 95% CI 2-sided [0.31 to 0.87] — Treatment comparison between placebo and nemiralisib 500 mcg at Day 84 was performed and posterior median odds ratio and 95% HPD CrI has been presented
Statistical Analysis 24: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 1.08, 95% CI 2-sided [0.73 to 1.47] — Treatment comparison between placebo and nemiralisib 750 mcg at Day 84 was performed and posterior median odds ratio and 95% HPD CrI has been presented

7. Secondary Outcome: Number of Participants With Time to Recovery From Index Exacerbation Using EXACT- PRO Tool
Description: Time to EXACT-defined recovery from index exacerbation is defined as time from the date of randomization until date of the first EXACT-defined recovery day during the 12-Week Treatment Period. EXACT-defined recovery from the index exacerbation is defined as a decrease in the Rolling Average EXACT total Score >=9 points from the Maximum Observed Value, sustained for >=7 days, with the first of the 7 days defined as the recovery day. Analysis was performed using a Bayesian Cox proportional hazards model adjusting for treatment group, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in the previous 12 months and gender. Number of participants reporting events is presented.
Time Frame: From randomization to Week 12
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants | 141 | 11 | 54 | 50 | 45 | 34 | 149
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median hazard ratio = 1.053, 95% CI 2-sided [0.477 to 1.765] — Treatment comparison between placebo and Nemiralisib 12.5 mcg was performed and posterior median hazard ratio and 95% HPD CrI has been presented
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median hazard ratio = 1.200, 95% CI 2-sided [0.840 to 1.597] — Treatment comparison between placebo and Nemiralisib 50 mcg was performed and posterior median hazard ratio and 95% HPD CrI has been presented
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median hazard ratio = 1.060, 95% CI 2-sided [0.734 to 1.432] — Treatment comparison between placebo and Nemiralisib 100 mcg was performed and posterior median hazard ratio and 95% HPD CrI has been presented
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median hazard ratio = 1.030, 95% CI 2-sided [0.719 to 1.413] — Treatment comparison between placebo and Nemiralisib 250 mcg was performed and posterior median hazard ratio and 95% HPD CrI has been presented
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median hazard ratio = 0.751, 95% CI 2-sided [0.487 to 1.057] — Treatment comparison between placebo and Nemiralisib 500 mcg was performed and posterior median hazard ratio and 95% HPD CrI has been presented
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median hazard ratio = 1.149, 95% CI 2-sided [0.899 to 1.426] — Treatment comparison between placebo and Nemiralisib 750 mcg was performed and posterior median hazard ratio and 95% HPD CrI has been presented

8. Secondary Outcome: Mean Severity of Subsequent Health Care Resource Use (HCRU) Exacerbations Defined by EXACT
Description: Severity of subsequent HCRU-defined exacerbations defined by EXACT was defined as the highest EXACT Total Score (not using the 3-day Rolling Average) during the period from date of onset of the subsequent HCRU-exacerbation until date of EXACT-defined recovery of subsequent exacerbation. EXACT-PRO, 14-item instrument to capture occurrence, frequency, severity, and duration of exacerbations using an eDiary. Total score ranges from 0-100, higher score indicates more severe condition. For participants with more than one subsequent exacerbation, severity was calculated for each subsequent exacerbation.
Time Frame: Up to Week 12
Population: Severity was derived for participants from MITT Population who had reported subsequent exacerbation. Only those participants with data available at specified data points were analyzed (represented by n=X in the category title).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 66 | 3 | 23 | 25 | 26 | 15 | 78
Scores on a scale
  Moderate/Severe, n=66, 3, 23, 25, 26, 15, 78 | 53.3 (12.16) | 64.6 (25.20) | 59.8 (12.82) | 50.5 (10.76) | 47.5 (13.95) | 57.6 (10.30) | 51.9 (10.78)
  Moderate, n=55, 3, 15, 23, 17, 10, 63: number analyzed (Participants) | 55 | 3 | 15 | 23 | 17 | 10 | 63
  Moderate, n=55, 3, 15, 23, 17, 10, 63 | 53.1 (11.54) | 60.0 (26.56) | 57.4 (11.08) | 50.0 (11.15) | 46.3 (14.20) | 53.8 (9.28) | 50.0 (10.17)
  Severe, n=13, 1, 9, 3, 10, 6, 20: number analyzed (Participants) | 13 | 1 | 9 | 3 | 10 | 6 | 20
  Severe, n=13, 1, 9, 3, 10, 6, 20 | 54.0 (15.53) | 83.0 (NA) — NA indicates standard deviation could not be calculated as only one participant was analyzed. | 64.0 (15.01) | 55.3 (5.69) | 49.5 (13.95) | 64.1 (8.99) | 58.8 (10.34)

9. Secondary Outcome: Percentage of Responders Using the COPD Assessment Test (CAT) on Treatment Days 28, 56, and 84, and Following EXACT Defined Recovery From the Index Exacerbation
Description: The CAT is a short, self-completed, 8-item questionnaire, each item was rated on a 6-point scale ranging from 0 (no impairment) to 5 (maximum impairment). The total CAT score is calculated by summing the scores of all items and ranges from 0 to 40, higher scores indicating severe condition. The percentage of responders using the CAT is defined as number of participants with a decrease from Baseline in CAT Total Score >=2 on or before Days 28, 56 and 84 divided by total number of participants in the MITT population. Percentage of responders using CAT was derived only for participants with a Baseline CAT Total Score >=2. Analysis was performed using a separate Bayesian logistic regression for each time point adjusting for treatment group, smoking status at baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in the previous 12 months and gender.
Time Frame: Days 28, 56 and 84
Population: MITT Population.
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Percentage of responders
  Day 28 | 32 | 36 | 34 | 39 | 38 | 34 | 25
  Day 56 | 63 | 50 | 73 | 61 | 69 | 55 | 61
  Day 84 | 70 | 55 | 78 | 65 | 72 | 60 | 66
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 1.22, 95% CI 2-sided [0.35 to 2.70] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.11, 95% CI 2-sided [0.63 to 1.77] — [estimate comment as in outcome 6, analysis 8]
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.41, 95% CI 2-sided [0.77 to 2.17] — [estimate comment as in outcome 6, analysis 9]
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.28, 95% CI 2-sided [0.71 to 2.00] — [estimate comment as in outcome 6, analysis 10]
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 1.11, 95% CI 2-sided [0.61 to 1.75] — [estimate comment as in outcome 6, analysis 11]
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 0.70, 95% CI 2-sided [0.46 to 0.99] — [estimate comment as in outcome 6, analysis 12]
Statistical Analysis 7: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 0.64, 95% CI 2-sided [0.20 to 1.41] — [estimate comment as in outcome 6, analysis 13]
Statistical Analysis 8: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.53, 95% CI 2-sided [0.84 to 2.46] — [estimate comment as in outcome 6, analysis 14]
Statistical Analysis 9: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 0.95, 95% CI 2-sided [0.53 to 1.48] — [estimate comment as in outcome 6, analysis 15]
Statistical Analysis 10: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.36, 95% CI 2-sided [0.74 to 2.16] — [estimate comment as in outcome 6, analysis 16]
Statistical Analysis 11: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.76, 95% CI 2-sided [0.43 to 1.17] — [estimate comment as in outcome 6, analysis 17]
Statistical Analysis 12: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 0.93, 95% CI 2-sided [0.63 to 1.27] — [estimate comment as in outcome 6, analysis 18]
Statistical Analysis 13: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 0.54, 95% CI 2-sided [0.16 to 1.20] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 14: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.53, 95% CI 2-sided [0.79 to 2.56] — [estimate comment as in outcome 6, analysis 20]
Statistical Analysis 15: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 0.83, 95% CI 2-sided [0.46 to 1.30] — [estimate comment as in outcome 6, analysis 21]
Statistical Analysis 16: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.16, 95% CI 2-sided [0.62 to 1.86] — [estimate comment as in outcome 6, analysis 22]
Statistical Analysis 17: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.65, 95% CI 2-sided [0.36 to 1.02] — [estimate comment as in outcome 6, analysis 23]
Statistical Analysis 18: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 0.85, 95% CI 2-sided [0.57 to 1.17] — [estimate comment as in outcome 6, analysis 24]

10. Secondary Outcome: Change From Baseline in CAT Total Score
Description: The CAT is a short, self-completed, 8-item questionnaire, each item was rated on a 6-point scale ranging from 0 (no impairment) to 5 (maximum impairment). The total CAT score was calculated by summing the scores of all items and ranges from 0 to 40, higher scores indicating more severe condition. Baseline (Day 1) is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in CAT Total Score is defined as CAT Total Score on Days 28, 56 and 84 minus Baseline CAT Total Score. Analysis was performed using Bayesian repeated measures model adjusting for Baseline by visit interaction, treatment by visit interaction, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in the previous 12 months and gender. Posterior adjusted median change from Baseline and 95% HPD CrI has been presented.
Time Frame: Baseline and at Days 28, 56 and 84
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Scores on a scale
  Day 28, n=234, 19, 86, 80, 77, 74, 229: number analyzed (Participants) | 234 | 19 | 86 | 80 | 77 | 74 | 229
  Day 28, n=234, 19, 86, 80, 77, 74, 229 | -4.7 [-5.6 to -3.8] | -2.3 [-5.1 to 0.5] | -4.0 [-5.4 to -2.7] | -3.9 [-5.4 to -2.4] | -5.1 [-6.5 to -3.7] | -3.1 [-4.5 to -1.6] | -4.7 [-5.6 to -3.8]
  Day 56, n=231, 20, 78, 77, 76, 69, 222: number analyzed (Participants) | 231 | 20 | 78 | 77 | 76 | 69 | 222
  Day 56, n=231, 20, 78, 77, 76, 69, 222 | -4.2 [-5.2 to -3.3] | -1.9 [-4.7 to 1.0] | -3.4 [-5.0 to -1.9] | -4.5 [-6.0 to -2.9] | -4.8 [-6.4 to -3.4] | -3.8 [-5.5 to -2.3] | -4.4 [-5.4 to -3.5]
  Day 84, n=218, 17, 75, 75, 69, 62, 213: number analyzed (Participants) | 218 | 17 | 75 | 75 | 69 | 62 | 213
  Day 84, n=218, 17, 75, 75, 69, 62, 213 | -4.6 [-5.6 to -3.6] | -2.7 [-6.0 to 0.3] | -3.5 [-5.0 to -1.9] | -5.1 [-6.7 to -3.5] | -4.7 [-6.3 to -3.1] | -3.8 [-5.4 to -2.1] | -4.2 [-5.2 to -3.2]
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = 2.4, 95% CI 2-sided [-0.5 to 5.2] — Treatment comparison between placebo and Nemiralisib 12.5 mcg at Day 28 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = 0.7, 95% CI 2-sided [-0.8 to 2.3] — Treatment comparison between placebo and Nemiralisib 50 mcg at Day 28 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = 0.8, 95% CI 2-sided [-0.8 to 2.4] — Treatment comparison between placebo and Nemiralisib 100 mcg at Day 28 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = -0.3, 95% CI 2-sided [-2.0 to 1.2] — Treatment comparison between placebo and Nemiralisib 250 mcg at Day 28 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjacent median difference = 1.6, 95% CI 2-sided [0.0 to 3.3] — Treatment comparison between placebo and Nemiralisib 500 mcg at Day 28 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = 0.0, 95% CI 2-sided [-1.1 to 1.1] — Treatment comparison between placebo and Nemiralisib 750 mcg at Day 28 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 7: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = 2.3, 95% CI 2-sided [-0.5 to 5.4] — Treatment comparison between placebo and Nemiralisib 12.5 mcg at Day 56 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 8: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = 0.8, 95% CI 2-sided [-0.9 to 2.4] — Treatment comparison between placebo and Nemiralisib 50 mcg at Day 56 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 9: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = -0.3, 95% CI 2-sided [-1.9 to 1.4] — Treatment comparison between placebo and Nemiralisib 100 mcg at Day 56 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 10: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = -0.5, 95% CI 2-sided [-2.3 to 1.0] — Treatment comparison between placebo and Nemiralisib 250 mcg at Day 56 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 11: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjusted median difference = 0.4, 95% CI 2-sided [-1.2 to 2.2] — Treatment comparison between placebo and Nemiralisib 500 mcg at Day 56 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 12: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = -0.2, 95% CI 2-sided [-1.4 to 1.0] — Treatment comparison between placebo and Nemiralisib 750 mcg at Day 56 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 13: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = 1.9, 95% CI 2-sided [-1.4 to 5.1] — Treatment comparison between placebo and Nemiralisib 12.5 mcg at Day 84 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 14: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = 1.1, 95% CI 2-sided [-0.7 to 2.8] — Treatment comparison between placebo and Nemiralisib 50 mcg at Day 84 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 15: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = -0.5, 95% CI 2-sided [-2.3 to 1.1] — Treatment comparison between placebo and Nemiralisib 100 mcg at Day 84 was performed and posterior adjsted median difference and 95% HPD CrI has been presented
Statistical Analysis 16: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = -0.1, 95% CI 2-sided [-1.9 to 1.7] — Treatment comparison between placebo and Nemiralisib 250 mcg at Day 84 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 17: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjusted median difference = 0.8, 95% CI 2-sided [-0.9 to 2.8] — Treatment comparison between placebo and Nemiralisib 500 mcg at Day 84 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 18: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = 0.4, 95% CI 2-sided [-0.8 to 1.7] — Treatment comparison between placebo and Nemiralisib 750 mcg at Day 84 was performed and posterior adjusted median difference and 95% HPD CrI has been presented

11. Secondary Outcome: Percentage of Responders on the St. George's Respiratory Questionnaire (SGRQ) Total Score as Measured by the SGRQ for COPD Participants (SGRQ-C) at Days 28, 56, and 84
Description: SGRQ-C is a 40-item questionnaire designed specifically to focus on COPD participants and was scored equivalent to the SGRQ Total Score, ranging from 0 to 100, where higher scores reflect worse health-related quality of life. The percentage of responders on the SGRQ Total Score was derived for participants with a Baseline SGRQ Total Score >=4. Percentage of responders on the SGRQ Total Score is defined as number of participants with a decrease from Baseline in SGRQ Total Score >=4 on or before Days 28, 56 and 84 divided by total number of participants in the MITT population. Analysis was performed using a separate Bayesian logistic regression for each time point adjusting for treatment group, smoking status at baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in the previous 12 months and gender.
Time Frame: Days 28, 56 and 84
Population: MITT Population.
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Percentage of responders
  Day 28: number analyzed (Participants) | 234 | 19 | 86 | 80 | 77 | 74 | 229
  Day 28 | 21 | 14 | 19 | 26 | 32 | 24 | 21
  Day 56: number analyzed (Participants) | 231 | 20 | 78 | 77 | 76 | 69 | 222
  Day 56 | 50 | 36 | 56 | 55 | 60 | 49 | 53
  Day 84: number analyzed (Participants) | 218 | 17 | 75 | 75 | 69 | 62 | 213
  Day 84 | 61 | 50 | 66 | 63 | 68 | 57 | 62
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 0.51, 95% CI 2-sided [0.03 to 1.41] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 0.87, 95% CI 2-sided [0.42 to 1.47] — [estimate comment as in outcome 6, analysis 8]
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.37, 95% CI 2-sided [0.69 to 2.24] — [estimate comment as in outcome 6, analysis 9]
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.78, 95% CI 2-sided [0.95 to 2.91] — [estimate comment as in outcome 6, analysis 10]
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 1.24, 95% CI 2-sided [0.61 to 2.08] — [estimate comment as in outcome 6, analysis 11]
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 0.95, 95% CI 2-sided [0.60 to 1.40] — [estimate comment as in outcome 6, analysis 12]
Statistical Analysis 7: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 0.54, 95% CI 2-sided [0.14 to 1.16] — [estimate comment as in outcome 6, analysis 13]
Statistical Analysis 8: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.27, 95% CI 2-sided [0.74 to 1.98] — [estimate comment as in outcome 6, analysis 14]
Statistical Analysis 9: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.29, 95% CI 2-sided [0.73 to 1.97] — [estimate comment as in outcome 6, analysis 15]
Statistical Analysis 10: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.47, 95% CI 2-sided [0.83 to 2.27] — [estimate comment as in outcome 6, analysis 16]
Statistical Analysis 11: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 1.04, 95% CI 2-sided [0.57 to 1.62] — [estimate comment as in outcome 6, analysis 17]
Statistical Analysis 12: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 1.10, 95% CI 2-sided [0.75 to 1.50] — [estimate comment as in outcome 6, analysis 18]
Statistical Analysis 13: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior median odds ratio = 0.63, 95% CI 2-sided [0.17 to 1.39] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 14: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior median odds ratio = 1.27, 95% CI 2-sided [0.72 to 2.01] — [estimate comment as in outcome 6, analysis 20]
Statistical Analysis 15: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior median odds ratio = 1.13, 95% CI 2-sided [0.64 to 1.79] — [estimate comment as in outcome 6, analysis 21]
Statistical Analysis 16: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior median odds ratio = 1.35, 95% CI 2-sided [0.75 to 2.14] — [estimate comment as in outcome 6, analysis 22]
Statistical Analysis 17: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior median odds ratio = 0.94, 95% CI 2-sided [0.53 to 1.45] — [estimate comment as in outcome 6, analysis 23]
Statistical Analysis 18: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior median odds ratio = 1.03, 95% CI 2-sided [0.71 to 1.43] — [estimate comment as in outcome 6, analysis 24]

12. Secondary Outcome: Change From Baseline in SGRQ Total Score at Days 28, 56 and 84
Description: SGRQ-C is a 40-item questionnaire designed specifically to focus on COPD participants and was scored equivalent to SGRQ Total Score, ranging from 0 to 100, where higher scores reflect worse health-related quality of life. Scores on a scale were calculated as 100 multiplied by summed weights from positive items in questionnaire divided by sum of weights of all items in questionnaire. Baseline (Day 1) is defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in SGRQ Total Score is defined as SGRQ Total Score on Days 28, 56 and 84 minus Baseline SGRQ Total Score. Analysis was performed using Bayesian repeated measures model adjusting for Baseline by visit interaction, treatment by visit interaction, smoking status at Baseline, region, severity of index exacerbation, number of moderate/severe exacerbations in previous 12 months and gender. Posterior adjusted median change from Baseline and 95% HPD CrI was presented
Time Frame: Baseline and Days 28, 56 and 84
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Scores on a scale
  Day 28, n=232, 19, 86, 78, 77, 72, 225: number analyzed (Participants) | 232 | 19 | 86 | 78 | 77 | 72 | 225
  Day 28, n=232, 19, 86, 78, 77, 72, 225 | -7.7 [-9.8 to -5.7] | -5.7 [-12.2 to 0.5] | -8.2 [-11.4 to -5.1] | -10.6 [-13.8 to -7.1] | -10.9 [-14.2 to -7.6] | -7.8 [-11.2 to -4.3] | -7.9 [-9.9 to -5.9]
  Day 56, n=227, 20, 78, 77, 74, 68, 219: number analyzed (Participants) | 227 | 20 | 78 | 77 | 74 | 68 | 219
  Day 56, n=227, 20, 78, 77, 74, 68, 219 | -8.0 [-10.2 to -6.0] | -3.9 [-10.4 to 2.8] | -9.3 [-12.5 to -5.9] | -10.7 [-14.1 to -7.3] | -11.3 [-14.6 to -7.6] | -8.9 [-12.6 to -5.5] | -8.4 [-10.6 to -6.3]
  Day 84, n=218, 17, 74, 74, 69, 60, 209: number analyzed (Participants) | 218 | 17 | 74 | 74 | 69 | 60 | 209
  Day 84, n=218, 17, 74, 74, 69, 60, 209 | -9.1 [-11.3 to -6.8] | -6.6 [-13.6 to 0.3] | -9.3 [-12.8 to -6.0] | -11.3 [-14.8 to -7.7] | -10.9 [-14.4 to -7.2] | -9.4 [-13.1 to -5.5] | -7.9 [-10.1 to -5.7]
Statistical Analysis 1: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = 2.0, 95% CI 2-sided [-4.8 to 8.3] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = -0.5, 95% CI 2-sided [-4.0 to 3.1] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = -2.9, 95% CI 2-sided [-6.2 to 1.1] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = -3.2, 95% CI 2-sided [-6.7 to 0.4] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjusted median difference = -0.1, 95% CI 2-sided [-4.0 to 3.5] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = -0.2, 95% CI 2-sided [-2.7 to 2.3] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = 4.1, 95% CI 2-sided [-2.5 to 11.0] — [estimate comment as in outcome 10, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = -1.2, 95% CI 2-sided [-4.8 to 2.5] — [estimate comment as in outcome 10, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = -2.7, 95% CI 2-sided [-6.3 to 1.1] — [estimate comment as in outcome 10, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = -3.3, 95% CI 2-sided [-7.3 to 0.4] — [estimate comment as in outcome 10, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjusted median difference = -0.8, 95% CI 2-sided [-4.6 to 3.0] — [estimate comment as in outcome 10, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = -0.4, 95% CI 2-sided [-2.9 to 2.5] — [estimate comment as in outcome 10, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs Nemiralisib 12.5 mcg; Test type: Other; Posterior adjusted median difference = 2.4, 95% CI 2-sided [-4.8 to 9.4] — [estimate comment as in outcome 10, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs Nemiralisib 50 mcg; Test type: Other; Posterior adjusted median difference = -0.2, 95% CI 2-sided [-4.1 to 3.6] — [estimate comment as in outcome 10, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs Nemiralisib 100 mcg; Test type: Other; Posterior adjusted median difference = -2.3, 95% CI 2-sided [-6.1 to 1.8] — Treatment comparison between placebo and Nemiralisib 100 mcg at Day 84 was performed and posterior adjusted median difference and 95% HPD CrI has been presented
Statistical Analysis 16: Comparison: Placebo vs Nemiralisib 250 mcg; Test type: Other; Posterior adjusted median difference = -1.8, 95% CI 2-sided [-5.7 to 2.3] — [estimate comment as in outcome 10, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs Nemiralisib 500 mcg; Test type: Other; Posterior adjusted median difference = -0.3, 95% CI 2-sided [-4.5 to 3.8] — [estimate comment as in outcome 10, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs Nemiralisib 750 mcg; Test type: Other; Posterior adjusted median difference = 1.2, 95% CI 2-sided [-1.7 to 4.0] — [estimate comment as in outcome 10, analysis 18]

13. Secondary Outcome: Mean Number of Occasions of Rescue Medication Use Per Day
Description: Albuterol (Salbutamol) MDI or nebules was used as a rescue medication. Rescue medication use was recorded as the number of occasions of rescue medication use each day. The mean number of occasions of rescue medication use per day is defined as sum of the number of occasions of rescue medication use each day within the time-period divided by the total number of days with non-missing values within the time-period. Over the 12-Week treatment period is defined as Day 1 to Day of last dose.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 of treatment and over the Week 12 treatment period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: No. of occasions of rescue use per day
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
No. of occasions of rescue use per day
  Week 1, n=254, 21, 87, 88, 80, 79, 254: number analyzed (Participants) | 254 | 21 | 87 | 88 | 80 | 79 | 254
  Week 1, n=254, 21, 87, 88, 80, 79, 254 | 1.699 (1.7674) | 2.112 (2.2977) | 1.633 (1.4320) | 1.926 (2.1569) | 1.670 (1.5728) | 1.917 (1.9298) | 1.747 (1.7332)
  Week 2, n=259, 21, 88, 89, 80, 82, 252: number analyzed (Participants) | 259 | 21 | 88 | 89 | 80 | 82 | 252
  Week 2, n=259, 21, 88, 89, 80, 82, 252 | 1.650 (1.8711) | 2.231 (2.7169) | 1.469 (1.4036) | 1.712 (2.0310) | 1.497 (1.5700) | 1.611 (1.7717) | 1.587 (1.6531)
  Week 3, n=256, 21, 90, 88, 80, 81, 245: number analyzed (Participants) | 256 | 21 | 90 | 88 | 80 | 81 | 245
  Week 3, n=256, 21, 90, 88, 80, 81, 245 | 1.729 (1.8157) | 2.021 (2.2926) | 1.495 (1.3943) | 1.693 (1.9679) | 1.488 (1.6611) | 1.742 (1.8380) | 1.655 (1.7430)
  Week 4, n=250, 21, 89, 87, 81, 77, 243: number analyzed (Participants) | 250 | 21 | 89 | 87 | 81 | 77 | 243
  Week 4, n=250, 21, 89, 87, 81, 77, 243 | 1.684 (1.7706) | 2.190 (2.3657) | 1.514 (1.5022) | 1.720 (2.0083) | 1.489 (1.6734) | 2.009 (2.0506) | 1.707 (1.7512)
  Week 5, n=251, 20, 88, 85, 78, 76, 240: number analyzed (Participants) | 251 | 20 | 88 | 85 | 78 | 76 | 240
  Week 5, n=251, 20, 88, 85, 78, 76, 240 | 1.735 (1.8662) | 2.329 (2.6394) | 1.533 (1.5706) | 1.750 (2.0380) | 1.535 (1.8384) | 1.949 (1.9685) | 1.737 (1.8030)
  Week 6, n=250, 20, 86, 84, 78, 72, 234: number analyzed (Participants) | 250 | 20 | 86 | 84 | 78 | 72 | 234
  Week 6, n=250, 20, 86, 84, 78, 72, 234 | 1.741 (1.9543) | 2.378 (2.6904) | 1.382 (1.4000) | 1.792 (2.0822) | 1.636 (1.8042) | 1.936 (2.0729) | 1.780 (1.8083)
  Week 7, n=250, 20, 85, 83, 77, 71, 231: number analyzed (Participants) | 250 | 20 | 85 | 83 | 77 | 71 | 231
  Week 7, n=250, 20, 85, 83, 77, 71, 231 | 1.703 (1.9914) | 2.479 (2.6976) | 1.531 (1.6374) | 1.697 (2.0769) | 1.628 (1.8741) | 1.899 (2.1694) | 1.826 (1.8778)
  Week 8, n=250, 20, 84, 83, 77, 71, 231: number analyzed (Participants) | 250 | 20 | 84 | 83 | 77 | 71 | 231
  Week 8, n=250, 20, 84, 83, 77, 71, 231 | 1.656 (1.8606) | 2.736 (3.1579) | 1.553 (1.5884) | 1.616 (1.9444) | 1.572 (1.8294) | 2.006 (2.2242) | 1.824 (1.8397)
  Week 9, n=244, 20, 82, 81, 76, 71, 229: number analyzed (Participants) | 244 | 20 | 82 | 81 | 76 | 71 | 229
  Week 9, n=244, 20, 82, 81, 76, 71, 229 | 1.708 (1.8709) | 2.765 (3.1104) | 1.608 (1.7699) | 1.658 (2.0646) | 1.720 (1.8918) | 1.953 (2.1838) | 1.775 (1.8753)
  Week 10, n=241, 20, 81, 80, 73, 71, 227: number analyzed (Participants) | 241 | 20 | 81 | 80 | 73 | 71 | 227
  Week 10, n=241, 20, 81, 80, 73, 71, 227 | 1.698 (1.9023) | 2.543 (2.8753) | 1.589 (1.6571) | 1.596 (1.9809) | 1.546 (1.8824) | 1.927 (2.1613) | 1.705 (1.7646)
  Week 11, n=241, 20, 79, 80, 73, 71, 226: number analyzed (Participants) | 241 | 20 | 79 | 80 | 73 | 71 | 226
  Week 11, n=241, 20, 79, 80, 73, 71, 226 | 1.729 (1.9406) | 2.164 (2.2504) | 1.404 (1.4897) | 1.602 (1.9435) | 1.672 (1.9447) | 1.926 (2.3243) | 1.716 (1.7421)
  Week 12, n=240, 20, 78, 80, 73, 70, 225: number analyzed (Participants) | 240 | 20 | 78 | 80 | 73 | 70 | 225
  Week 12, n=240, 20, 78, 80, 73, 70, 225 | 1.666 (1.7913) | 2.386 (2.8157) | 1.414 (1.3920) | 1.671 (1.9612) | 1.712 (1.9532) | 1.790 (2.1140) | 1.731 (1.7245)
  Over 12 Week, n=273, 21, 91, 91, 86, 83, 268: number analyzed (Participants) | 273 | 21 | 91 | 91 | 86 | 83 | 268
  Over 12 Week, n=273, 21, 91, 91, 86, 83, 268 | 1.684 (1.6903) | 2.330 (2.4715) | 1.553 (1.4044) | 1.750 (1.9048) | 1.620 (1.5994) | 1.921 (1.9201) | 1.733 (1.6618)

14. Secondary Outcome: Percentage of Rescue-free Days
Description: Albuterol (Salbutamol) MDI or nebules was used as a rescue medication. Percentage of Rescue-Free Days is defined as sum of the number of days where the number of occasions of rescue medication use is zero within the time-period divided by total number of days with non-missing values within the time-period multiplied by 100 where the time-period is defined as follows: Week 1: Day 1-7; Week 2: Day 8 - 14; Week 3: Day 15-21; Week 4: Day 22-28; Week 5: Day 29-35; Week 6: Day 36-42; Week 7: Day 43-49; Week 8: Day 50-56; Week 9: Day 57-63; Week 10: Day 64-70; Week 11: Day 71-77; Week 12: Day 78 to Day of last dose; Over the 12-Week: Day 1 to Day of last dose.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 of treatment and over the Week 12 treatment period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of rescue free days
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Percentage of rescue free days
  Week 1, n=254, 21, 87, 88, 80, 79, 254: number analyzed (Participants) | 254 | 21 | 87 | 88 | 80 | 79 | 254
  Week 1, n=254, 21, 87, 88, 80, 79, 254 | 34.898 (37.7118) | 36.076 (44.3182) | 29.849 (38.3385) | 33.392 (39.7372) | 32.583 (38.3577) | 34.453 (35.9802) | 29.779 (36.1498)
  Week 2, n=259, 21, 88, 89, 80, 82, 252: number analyzed (Participants) | 259 | 21 | 88 | 89 | 80 | 82 | 252
  Week 2, n=259, 21, 88, 89, 80, 82, 252 | 41.002 (40.9566) | 40.819 (46.7899) | 32.145 (41.2227) | 43.017 (43.9884) | 38.573 (40.3629) | 40.595 (41.1717) | 33.639 (38.9767)
  Week 3, n=256, 21, 90, 88, 80, 81, 245: number analyzed (Participants) | 256 | 21 | 90 | 88 | 80 | 81 | 245
  Week 3, n=256, 21, 90, 88, 80, 81, 245 | 38.204 (39.0621) | 38.776 (44.0612) | 31.643 (38.0943) | 39.964 (40.3936) | 41.191 (42.1751) | 34.923 (40.4026) | 33.006 (38.4986)
  Week 4, n=250, 21, 89, 87, 81, 77, 243: number analyzed (Participants) | 250 | 21 | 89 | 87 | 81 | 77 | 243
  Week 4, n=250, 21, 89, 87, 81, 77, 243 | 39.678 (40.8359) | 35.376 (43.9405) | 32.531 (39.0078) | 42.202 (43.0692) | 43.194 (41.0201) | 30.986 (38.5941) | 32.394 (39.0174)
  Week 5, n=251, 20, 88, 85, 78, 76, 240: number analyzed (Participants) | 251 | 20 | 88 | 85 | 78 | 76 | 240
  Week 5, n=251, 20, 88, 85, 78, 76, 240 | 38.262 (40.7807) | 35.005 (41.8344) | 35.552 (40.5745) | 41.682 (41.3648) | 41.026 (42.1584) | 33.912 (37.9973) | 33.168 (39.0654)
  Week 6, n=250, 20, 86, 84, 78, 72, 234: number analyzed (Participants) | 250 | 20 | 86 | 84 | 78 | 72 | 234
  Week 6, n=250, 20, 86, 84, 78, 72, 234 | 40.287 (42.2167) | 37.870 (40.2125) | 35.384 (40.9175) | 41.720 (44.0117) | 39.196 (41.6575) | 35.519 (42.2122) | 32.351 (39.2542)
  Week 7, n=250, 20, 85, 83, 77, 71, 231: number analyzed (Participants) | 250 | 20 | 85 | 83 | 77 | 71 | 231
  Week 7, n=250, 20, 85, 83, 77, 71, 231 | 41.373 (43.4266) | 32.145 (43.1992) | 35.634 (41.3319) | 45.266 (43.5910) | 40.409 (42.0560) | 38.232 (41.0296) | 31.975 (39.4910)
  Week 8, n=250, 20, 84, 83, 77, 71, 231: number analyzed (Participants) | 250 | 20 | 84 | 83 | 77 | 71 | 231
  Week 8, n=250, 20, 84, 83, 77, 71, 231 | 42.058 (41.2168) | 34.290 (42.8300) | 33.029 (41.0867) | 44.118 (41.6682) | 42.918 (42.8354) | 34.811 (39.3585) | 32.357 (39.9221)
  Week 9, n=244, 20, 82, 81, 76, 71, 229: number analyzed (Participants) | 244 | 20 | 82 | 81 | 76 | 71 | 229
  Week 9, n=244, 20, 82, 81, 76, 71, 229 | 39.268 (40.5300) | 32.145 (44.6657) | 32.759 (39.2972) | 42.505 (41.2121) | 39.476 (42.2376) | 36.823 (42.3513) | 33.606 (39.4690)
  Week 10, n=241, 20, 81, 80, 73, 71, 227: number analyzed (Participants) | 241 | 20 | 81 | 80 | 73 | 71 | 227
  Week 10, n=241, 20, 81, 80, 73, 71, 227 | 40.608 (41.0492) | 35.000 (42.3430) | 32.456 (40.7192) | 43.396 (42.3040) | 41.492 (42.1984) | 37.024 (41.2291) | 33.483 (40.1924)
  Week 11, n=241, 20, 79, 80, 73, 71, 226: number analyzed (Participants) | 241 | 20 | 79 | 80 | 73 | 71 | 226
  Week 11, n=241, 20, 79, 80, 73, 71, 226 | 39.701 (41.9689) | 38.575 (44.2366) | 35.624 (42.6625) | 42.859 (41.7845) | 39.337 (42.3061) | 39.841 (43.7237) | 33.127 (39.1842)
  Week 12, n=240, 20, 78, 80, 73, 70, 225: number analyzed (Participants) | 240 | 20 | 78 | 80 | 73 | 70 | 225
  Week 12, n=240, 20, 78, 80, 73, 70, 225 | 41.390 (40.8871) | 39.415 (45.0442) | 37.369 (40.2613) | 41.300 (39.8199) | 39.981 (40.8296) | 42.236 (42.1567) | 33.906 (38.4851)
  Over 12 Week, n=273, 21, 91, 91, 86, 83, 268: number analyzed (Participants) | 273 | 21 | 91 | 91 | 86 | 83 | 268
  Over 12 Week, n=273, 21, 91, 91, 86, 83, 268 | 39.743 (36.8957) | 35.533 (39.0694) | 33.590 (36.6456) | 40.441 (37.6285) | 39.631 (36.5157) | 35.820 (34.6377) | 32.743 (33.9362)

15. Secondary Outcome: Plasma Concentration of Nemiralisib
Description: Plasma samples were collected at indicated time points and analyzed for concentrations of Nemiralisb. Pharmacokinetic (PK) Population consists of all participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). Participants were summarized according to the treatment that they actually received.
Time Frame: Pre-dose, 0-1 hour, >1-6 hours post-dose on Days 14 and 28
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 5 | 22 | 24 | 19 | 20 | 73
Picograms per milliliter
  Day 14, Pre-dose, n=2, 19, 24, 16, 18, 69: number analyzed (Participants) | 2 | 19 | 24 | 16 | 18 | 69
  Day 14, Pre-dose, n=2, 19, 24, 16, 18, 69 | 113.6 (6) | 62.0 (46) | 142.8 (44) | 416.0 (59) | 687.3 (53) | 1069.6 (70)
  Day 14, 0-1 hour, n=4, 19, 24, 15, 18, 67: number analyzed (Participants) | 4 | 19 | 24 | 15 | 18 | 67
  Day 14, 0-1 hour, n=4, 19, 24, 15, 18, 67 | 54.9 (43) | 109.9 (51) | 253.7 (73) | 767.6 (71) | 1492.0 (59) | 1972.0 (110)
  Day 14, >1-6 hours, n=4, 20, 23, 15, 18, 65: number analyzed (Participants) | 4 | 20 | 23 | 15 | 18 | 65
  Day 14, >1-6 hours, n=4, 20, 23, 15, 18, 65 | 35.0 (57) | 93.1 (58) | 231.8 (53) | 657.0 (61) | 1146.7 (56) | 1622.7 (90)
  Day 28, Pre-dose, n=2, 18, 23, 16, 16, 67: number analyzed (Participants) | 2 | 18 | 23 | 16 | 16 | 67
  Day 28, Pre-dose, n=2, 18, 23, 16, 16, 67 | 23.6 (24) | 60.5 (45) | 129.4 (46) | 315.6 (85) | 528.3 (110) | 937.6 (101)
  Day 28, 0-1 hour, n=3, 19, 23, 16, 15, 63: number analyzed (Participants) | 3 | 19 | 23 | 16 | 15 | 63
  Day 28, 0-1 hour, n=3, 19, 23, 16, 15, 63 | 36.2 (26) | 104.9 (70) | 253.3 (52) | 807.0 (66) | 1552.2 (83) | 1717.6 (114)
  Day 28, >1-6 hours, n=3, 18, 23, 16, 14, 64: number analyzed (Participants) | 3 | 18 | 23 | 16 | 14 | 64
  Day 28, >1-6 hours, n=3, 18, 23, 16, 14, 64 | 28.1 (15) | 85.4 (40) | 211.4 (41) | 598.8 (39) | 1079.5 (80) | 1388.1 (101)

16. Other Pre Specified Outcome: Area Under the Concentration Time Curve (AUC) From Time Zero to 24 Hours [AUC(0-24)] of Nemiralisib
Description: Plasma samples were collected at indicated time points and analyzed.
Time Frame: Pre-dose, 0-1 hour, >1-6 hours post-dose on Days 14 and 28
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms per milliliter
Arm/Group | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 5 | 22 | 24 | 19 | 20 | 73
Hours*picograms per milliliter | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary population pharmacokinetic (Pop PK) analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted

17. Other Pre Specified Outcome: AUC From Time Zero to Time 't' [AUC(0-t)] of Nemiralisib
Description: Plasma samples were collected at indicated time points and analyzed.
Time Frame: Pre-dose, 0-1 hour, >1-6 hours post-dose on Days 14 and 28
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms per milliliter
Arm/Group | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 5 | 22 | 24 | 19 | 20 | 73
Hours*picograms per milliliter | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted

18. Other Pre Specified Outcome: Maximum Observed Plasma Drug Concentration (Cmax) of Nemiralisib
Description: Plasma samples were collected at indicated time points and analyzed.
Time Frame: Pre-dose, 0-1 hour, >1-6 hours post-dose on Days 14 and 28
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 5 | 22 | 24 | 19 | 20 | 73
Picograms per milliliter | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted

19. Other Pre Specified Outcome: Time to Reach Cmax (Tmax) of Nemiralisib
Description: Plasma samples were collected at indicated time points and analyzed.
Time Frame: Pre-dose, 0-1 hour, >1-6 hours post-dose on Days 14 and 28
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 5 | 22 | 24 | 19 | 20 | 73
Hours | NA [NA to NA] — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA [NA to NA] — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA [NA to NA] — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA [NA to NA] — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA [NA to NA] — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA [NA to NA] — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted

20. Other Pre Specified Outcome: Plasma Drug Concentration at Pre-dose (Ctrough) of Nemiralisib
Description: Plasma samples were collected at indicated time points and analyzed.
Time Frame: Pre-dose, 0-1 hour, >1-6 hours post-dose on Days 14 and 28
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 5 | 22 | 24 | 19 | 20 | 73
Picograms per milliliter | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted | NA (NA) — This was a conditional secondary endpoint for which results are not available because development of the associated asset was terminated and therefore secondary Pop PK analyses were not conducted

21. Secondary Outcome: Number of Participants Reporting Non-serious Adverse Events (Non-SAEs), SAEs and AE of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect and other important medical events. Safety Population consists of all randomized participants who received at least one dose of study treatment. Participants were summarized according to treatment that they actually received.
Time Frame: Up to Week 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants
  Any non-SAE | 31 | 1 | 14 | 19 | 25 | 36 | 101
  Any SAE | 23 | 2 | 9 | 13 | 16 | 6 | 26
  Any AESI | 9 | 0 | 10 | 10 | 21 | 29 | 93

22. Secondary Outcome: Number of Participants With Worst Case Post Baseline Diastolic Blood Pressure (DBP), Systolic Blood Pressure (SBP) and Pulse Rate
Description: The DBP, SBP and pulse rate were measured with participants seated at least 5 minutes before the assessments. Participants are counted in the worst case category if their value changes to (low, within range or no change, or high). Participants whose value category was unchanged (e.g., High to High), or whose value became within range, are recorded in the "To w/in Range or No Change" category. Participants are counted twice if the participant has values that changed "To Low" and "To High", so the percentages may not add to 100%. Participants with missing baseline value are assumed to have within range value.
Time Frame: Up to Week 16
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 271 | 21 | 91 | 92 | 88 | 88 | 266
Participants
  DBP, To low | 8 | 3 | 3 | 0 | 4 | 4 | 7
  DBP, To within range/no change | 260 | 17 | 85 | 91 | 79 | 82 | 256
  DBP, To high | 3 | 1 | 3 | 1 | 5 | 2 | 3
  Pulse rate, To low | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate,To within range/no change | 265 | 21 | 84 | 90 | 82 | 83 | 258
  Pulse rate, To high | 5 | 0 | 7 | 2 | 6 | 5 | 8
  SBP, To low | 11 | 1 | 5 | 3 | 2 | 3 | 8
  SBP, To withinn range/no change | 250 | 18 | 83 | 82 | 79 | 80 | 239
  SBP, To high | 10 | 2 | 3 | 7 | 8 | 6 | 19

23. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: A single 12-lead ECG with a 15-second rhythm strip was obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT and corrected QT (QTc) intervals. Abnormal ECG findings are presented.
Time Frame: Screening, Days 14, 84, 112 and at early withdrawal
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants
  Screening | 93 | 10 | 25 | 37 | 28 | 21 | 86
  Day 14 | 88 | 8 | 24 | 33 | 29 | 18 | 74
  Day 84 | 79 | 8 | 22 | 27 | 24 | 18 | 64
  Day 112 | 77 | 11 | 28 | 28 | 25 | 20 | 75
  Early withdrawal | 3 | 0 | 2 | 1 | 3 | 1 | 4

24. Secondary Outcome: Number of Participants With Worst Case Post Baseline Clinical Chemistry Values
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: blood urea nitrogen (BUN), creatinine (Crt), glucose (Glu), potassium (Pot), sodium (Sod), calcium (Cal), aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total and direct bilirubin, total protein and albumin (Alb). Participants are counted in the worst case category if their value changes to (low, within range or no change, or high). Participants whose value category was unchanged (e.g., High to High), or whose value became within range, are recorded in the "To w/in Range or No Change" category. Participants are counted twice if the participant has values that changed "To Low" and "To High", so the percentages may not add to 100%. Participants with missing baseline value are assumed to have within range value.
Time Frame: Upto Week 16
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants
  Alb,To low, n=266, 21, 91, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Alb,To low, n=266, 21, 91, 90, 87, 85, 263 | 2 | 0 | 0 | 0 | 1 | 1 | 2
  Alb,w/in range/no change,n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Alb,w/in range/no change,n=266,21,91,90,87,85,263 | 264 | 21 | 90 | 90 | 85 | 84 | 261
  Alb,To high,n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Alb,To high,n=266,21,91,90,87,85,263 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Cal,To low, n=266, 21, 90, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 90 | 90 | 87 | 85 | 263
  Cal,To low, n=266, 21, 90, 90, 87, 85, 263 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Cal,w/in range/no change,n=266,21,90,90,87,85,263: number analyzed (Participants) | 266 | 21 | 90 | 90 | 87 | 85 | 263
  Cal,w/in range/no change,n=266,21,90,90,87,85,263 | 265 | 21 | 90 | 90 | 87 | 84 | 262
  Cal,To high, n=266,21,90,90,87,85,263: number analyzed (Participants) | 266 | 21 | 90 | 90 | 87 | 85 | 263
  Cal,To high, n=266,21,90,90,87,85,263 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Crt,To low, n=266, 21, 91, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Crt,To low, n=266, 21, 91, 90, 87, 85, 263 | 27 | 3 | 10 | 7 | 4 | 9 | 32
  Crt,w/in range/no change,n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Crt,w/in range/no change,n=266,21,91,90,87,85,263 | 237 | 18 | 81 | 82 | 80 | 76 | 231
  Crt,To high, n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Crt,To high, n=266,21,91,90,87,85,263 | 2 | 0 | 0 | 1 | 3 | 0 | 0
  Glu,To low, n=266, 21, 91, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Glu,To low, n=266, 21, 91, 90, 87, 85, 263 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Glu,w/in range/no change,n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Glu,w/in range/no change,n=266,21,91,90,87,85,263 | 266 | 21 | 91 | 89 | 87 | 85 | 263
  Glu,To high, n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Glu,To high, n=266,21,91,90,87,85,263 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,To low, n=266, 21, 90, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 90 | 90 | 87 | 85 | 263
  Pot,To low, n=266, 21, 90, 90, 87, 85, 263 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,w/in range/no change,n=266,21,90,90,87,85,263: number analyzed (Participants) | 266 | 21 | 90 | 90 | 87 | 85 | 263
  Pot,w/in range/no change,n=266,21,90,90,87,85,263 | 264 | 21 | 90 | 90 | 86 | 84 | 262
  Pot,To high, n=266,21,90,90,87,85,263: number analyzed (Participants) | 266 | 21 | 90 | 90 | 87 | 85 | 263
  Pot,To high, n=266,21,90,90,87,85,263 | 2 | 0 | 0 | 0 | 1 | 1 | 1
  Sod,To low, n=266, 21, 91, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Sod,To low, n=266, 21, 91, 90, 87, 85, 263 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sod,w/in range/no change,n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Sod,w/in range/no change,n=266,21,91,90,87,85,263 | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Sod,To high, n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  Sod,To high, n=266,21,91,90,87,85,263 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN,To low, n=266, 21, 91, 90, 87, 85, 263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  BUN,To low, n=266, 21, 91, 90, 87, 85, 263 | 7 | 0 | 3 | 2 | 2 | 3 | 6
  BUN,w/in range/no change,n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  BUN,w/in range/no change,n=266,21,91,90,87,85,263 | 256 | 21 | 88 | 86 | 85 | 82 | 253
  BUN,To high, n=266,21,91,90,87,85,263: number analyzed (Participants) | 266 | 21 | 91 | 90 | 87 | 85 | 263
  BUN,To high, n=266,21,91,90,87,85,263 | 3 | 0 | 0 | 2 | 0 | 0 | 4

25. Secondary Outcome: Number of Participants With Worst Case Post Baseline Hematology Values
Description: Blood samples were collected for the analysis of hematology parameters including: platelets (Pla), red blood cells count, Hemoglobin (Hb), Hematocrit, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), percentage reticulocytes, neutrophils (Neu), lymphocytes (Lym), monocytes, eosinophils, leukocytes (Leu) and basophils. Participants are counted in the worst case category if their value changes to (low, within range or no change, or high). Participants whose value category was unchanged (e.g., High to High), or whose value became within range, are recorded in the "To w/in Range or No Change" category. Participants are counted twice if the participant has values that changed "To Low" and "To High", so the percentages may not add to 100%. Participants with missing baseline value are assumed to have within range value.
Time Frame: Upto Week 16
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants
  Hb,To low, n=260, 20, 90, 90, 84, 81, 254: number analyzed (Participants) | 260 | 20 | 90 | 90 | 84 | 81 | 254
  Hb,To low, n=260, 20, 90, 90, 84, 81, 254 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hb,w/in range/no change,n=260,20,90,90,84,81,254: number analyzed (Participants) | 260 | 20 | 90 | 90 | 84 | 81 | 254
  Hb,w/in range/no change,n=260,20,90,90,84,81,254 | 260 | 20 | 90 | 90 | 84 | 81 | 253
  Hb,To high,n=260, 20, 90, 90, 84, 81, 254: number analyzed (Participants) | 260 | 20 | 90 | 90 | 84 | 81 | 254
  Hb,To high,n=260, 20, 90, 90, 84, 81, 254 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Leu,To low,n=259, 20, 90, 90, 83, 78, 251: number analyzed (Participants) | 259 | 20 | 90 | 90 | 83 | 78 | 251
  Leu,To low,n=259, 20, 90, 90, 83, 78, 251 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leu,w/in range/no change,n=259,20,90,90,83,78,251: number analyzed (Participants) | 259 | 20 | 90 | 90 | 83 | 78 | 251
  Leu,w/in range/no change,n=259,20,90,90,83,78,251 | 211 | 16 | 81 | 74 | 63 | 62 | 201
  Leu,To high, n=259,20,90,90,83,78,251: number analyzed (Participants) | 259 | 20 | 90 | 90 | 83 | 78 | 251
  Leu,To high, n=259,20,90,90,83,78,251 | 48 | 4 | 9 | 16 | 20 | 16 | 50
  Lym,To low, n=256, 20, 85, 88, 82, 77, 249: number analyzed (Participants) | 256 | 20 | 85 | 88 | 82 | 77 | 249
  Lym,To low, n=256, 20, 85, 88, 82, 77, 249 | 8 | 1 | 6 | 7 | 7 | 2 | 11
  Lym,w/in range/no change,n=256,20,85,88,82,77,249: number analyzed (Participants) | 256 | 20 | 85 | 88 | 82 | 77 | 249
  Lym,w/in range/no change,n=256,20,85,88,82,77,249 | 239 | 19 | 79 | 76 | 70 | 73 | 226
  Lym,To high,n=256,20,85,88,82,77,249: number analyzed (Participants) | 256 | 20 | 85 | 88 | 82 | 77 | 249
  Lym,To high,n=256,20,85,88,82,77,249 | 9 | 0 | 0 | 5 | 5 | 2 | 12
  Neu, To low, n=256,20,85,88,82,77,249: number analyzed (Participants) | 256 | 20 | 85 | 88 | 82 | 77 | 249
  Neu, To low, n=256,20,85,88,82,77,249 | 3 | 0 | 1 | 1 | 0 | 0 | 2
  Neu,w/in range/no change,n=256,20,85,88,82,77,249: number analyzed (Participants) | 256 | 20 | 85 | 88 | 82 | 77 | 249
  Neu,w/in range/no change,n=256,20,85,88,82,77,249 | 215 | 17 | 73 | 76 | 68 | 60 | 213
  Neu,To high, n=256,20,85,88,82,77,249: number analyzed (Participants) | 256 | 20 | 85 | 88 | 82 | 77 | 249
  Neu,To high, n=256,20,85,88,82,77,249 | 38 | 3 | 11 | 11 | 14 | 17 | 34
  Pla,To low, n=253, 19, 88, 90, 84, 78, 245: number analyzed (Participants) | 253 | 19 | 88 | 90 | 84 | 78 | 245
  Pla,To low, n=253, 19, 88, 90, 84, 78, 245 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pla,w/in range/no change,n=253,19,88,90,84,78,245: number analyzed (Participants) | 253 | 19 | 88 | 90 | 84 | 78 | 245
  Pla,w/in range/no change,n=253,19,88,90,84,78,245 | 253 | 19 | 88 | 90 | 84 | 78 | 245
  Pla,To high, n=253,19,88,90,84,78,245: number analyzed (Participants) | 253 | 19 | 88 | 90 | 84 | 78 | 245
  Pla,To high, n=253,19,88,90,84,78,245 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants Reporting COPD Exacerbations
Description: Participants reporting acute COPD exacerbations during the study period has been presented.
Time Frame: Up to Week 16
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
Number analyzed (Participants) | 276 | 22 | 91 | 92 | 90 | 89 | 278
Participants | 8 | 1 | 6 | 4 | 4 | 3 | 17

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to Week 24
Description: Non-serious AEs and SAEs were summarized for the Safety Population.
Arm/Group | Placebo | Nemiralisib 12.5 mcg | Nemiralisib 50 mcg | Nemiralisib 100 mcg | Nemiralisib 250 mcg | Nemiralisib 500 mcg | Nemiralisib 750 mcg
All-Cause Mortality (participants affected / at risk) | 1/276 | 0/22 | 3/91 | 1/92 | 0/90 | 0/89 | 1/278
Serious Adverse Events (participants affected / at risk) | 23/276 | 2/22 | 9/91 | 13/92 | 16/90 | 6/89 | 26/278
Other Adverse Events (participants affected / at risk) | 31/276 | 1/22 | 14/91 | 19/92 | 25/90 | 36/89 | 101/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=276) | Nemiralisib 12.5 mcg (N=22) | Nemiralisib 50 mcg (N=91) | Nemiralisib 100 mcg (N=92) | Nemiralisib 250 mcg (N=90) | Nemiralisib 500 mcg (N=89) | Nemiralisib 750 mcg (N=278)
Chroni obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 6 (7) | 4 (4) | 4 (5) | 3 (3) | 17 (17)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=276) | Nemiralisib 12.5 mcg (N=22) | Nemiralisib 50 mcg (N=91) | Nemiralisib 100 mcg (N=92) | Nemiralisib 250 mcg (N=90) | Nemiralisib 500 mcg (N=89) | Nemiralisib 750 mcg (N=278)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0) | 10 (12) | 11 (17) | 23 (27) | 31 (58) | 96 (141)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 23 (41) | 1 (1) | 6 (8) | 8 (10) | 4 (5) | 2 (2) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03345407/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03345407/SAP_001.pdf